CLINICAL TRIAL: NCT01889992
Title: Cardiac Allograft Remodeling and Effects of Sirolimus on Its Progression
Brief Title: Cardiac Allograft Remodeling and Effects of Sirolimus
Acronym: CAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left University and project not continued
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0339-12-FB
Record Dates: First submitted 2013-06-19; First posted 2013-07-01 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Hypertrophy; Immunosuppression
Keywords: Heart transplantation; Cardiac allograft remodeling; Immunosuppression; Cardiac MRI; M-TOR inhibitor
MeSH Terms: conditions — Cardiomegaly | interventions — Sirolimus; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cardiac biopsy C4D stain (Active Comparator): A procedure that removes a very small sample of your heart muscle so that it can be evaluated in the lab. This procedure may be done to determine the cause of cardiac myopathy (a weakened heart muscle) or to check for rejection after a heart transplant.
  Interventions: Procedure: Cardiac Biopsy C4D stain
- Genetic Mechanism of M-TOR (Experimental): To identify the molecular and genetic mechanisms associated with development of early post-transplant CAR, and to evaluate the impact of mTOR-inhibitor Sirolimus on this process.
  Sirolimus dosage is based on blood levels.
  Interventions: Genetic: Genetic Mechanism of M-TOR
- Cardiac MRI (Active Comparator): Cardiac Magnetic Resonance Imaging (MRI) produces no side effects from the magnetic fields and radio waves and doesn't carry a risk of cancer or birth defects. Serious reactions to the special contrast dyes used for MRI are very rare. The MRI examination poses almost no risk to the average patient when appropriate safety guidelines are followed, however side effects are possible and include headache, nausea, dizziness, change in taste and allergic reaction. Such reactions usually are mild and easily controlled by medication.
  Interventions: Radiation: Cardiac MRI
- Coronary Angiography with IVUS (Active Comparator): Coronary angiography is a test that uses dye and special x rays to show the insides of your coronary arteries. The coronary arteries supply oxygen-rich blood to your heart.
  Intravascular ultrasound is a test that uses sound waves to see inside blood vessels. This article discusses intravascular ultrasound to see inside the coronary arteries, the blood vessels that supply the heart.
  Interventions: Procedure: Coronary angiography with IVUS
- Cardiopulmonary Exercise Test (CPET) (Active Comparator): Is a highly sensitive, non-invasive stress test. It is considered a stress test because the exercise stresses your body's systems by making them work faster and harder. A disease or condition that affects the heart, lungs or muscles will limit how much faster and harder these systems can work. A CPET assesses how well the heart, lungs, and muscles are working individually, and how these systems are working in unison. Your heart and lungs work together to deliver oxygen to your muscles, where it is used to make energy, and to remove carbon dioxide from your body.
  Interventions: Other: Cardiopulmonary Exercise Test (CPET)
- MTor Immunosuppression (Experimental): Sirolimus
  Sirolimus dosage is based on blood levels.
  To assess the potential of mTOR immunosuppressant Sirolimus in attenuation of CAR in HTx recipients and therefore, improve pre-existing cardiac allograft function, vasculopathy, and exercise capacity.
  Interventions: Radiation: Cardiac MRI; Procedure: Coronary angiography with IVUS; Other: Cardiac Allograft Remodeling; Drug: M-TOR Immunosuppression
- Cardiac Allograft Remodeling (Experimental): A surgical procedure in wich a diseased heart is replaced with a healthy heart from a deceased person.
  Interventions: Other: Cardiac Allograft Remodeling

INTERVENTIONS:
Radiation: Cardiac MRI — 1 month post HTx, year 1 and year 2 annual post HTx eval. CMRIs completed using 1.5-Tesla Whole Body MRI system. Scout images will determine short & long-axis views of the heart. ECG-gated cine MR of 3 long axis and a contiguous short axis orientation will be obtained. T1-weighted delayed enhancement images will be obtained 10 minutes after injection of a gadolinium-based contrast agent. Measurements from each slice will be summed using the method of disks. Myocardial mass will be estimated by multiplying the myocardial wall volume at end diastole by the specific gravity of muscle (1.05gm/ml) and LV hypertrophy will be defined as LV mass indexed to height in meters 2.7 >/=35.8 g/m 2.7) (18). Delayed Gadolinium enhancement will be defined as any enhancement pattern greater than 0%.
  Arms: Cardiac MRI; MTor Immunosuppression
Procedure: Coronary angiography with IVUS — Coronary angiography is a test that uses dye and special x rays to show the insides of your coronary arteries. The coronary arteries supply oxygen-rich blood to your heart.
  Intravascular ultrasound is a test that uses sound waves to see inside blood vessels. This article discusses intravascular ultrasound to see inside the coronary arteries, the blood vessels that supply the heart.
  Arms: Coronary Angiography with IVUS; MTor Immunosuppression
Other: Cardiac Allograft Remodeling — A surgical procedure in which a diseased heart is replaced with a healthy heart from a deceased person.
  Other Names: heart hypertrophy
  Arms: Cardiac Allograft Remodeling; MTor Immunosuppression
Drug: M-TOR Immunosuppression — Sirolimus (INN/USAN), also known as rapamycin, is an immunosuppressant drug used to prevent rejection in organ transplantation; it is especially useful in kidney transplants. It prevents activation of T cells and B-cells by inhibiting their response to interleukin-2 (IL-2).
  Sirolimus dosage based on blood levels.
  Other Names: Sirolimus
  Arms: MTor Immunosuppression
Procedure: Cardiac Biopsy C4D stain — A long, thin tube called a biopsy catheter is inserted through a vein in your neck or grion and guided through your blood vessels to your heart.
  Other Names: heart biopsy
  Arms: Cardiac biopsy C4D stain
Genetic: Genetic Mechanism of M-TOR — To identify the molecular and genetic mechanisms associated with development of early post-transplant CAR, and to evaluate the impact of mTOR-inhibitor Sirolimus on this process.
  Arms: Genetic Mechanism of M-TOR
Other: Cardiopulmonary Exercise Test (CPET) — The Cardiopulmonary Exercise Test is a highly sensitive, non-invasive stress test. It is considered a stress test because the exercise stresses your body's systems by making them work faster and harder. A disease or condition that affects the heart, lungs or muscles will limit how much faster and harder these systems can work. A CPET assesses how well the heart, lungs, and muscles are working individually, and how these systems are working in unison. Your heart and lungs work together to deliver oxygen to your muscles, where it is used to make energy, and to remove carbon dioxide from your body.
  Other Names: Stress test
  Arms: Cardiopulmonary Exercise Test (CPET)

SUMMARY:
Cardiac allograft remodeling causes poor quality of life, allograft failure and increased mortality after heart transplantation. Risk factors for cardiac allograft remodeling and its progression are poorly defined and there is a need for effective interventions.This is a multi-factorial phenomenon, associated with various immunological and non-immunological factors. Animal studies suggest M-TOR inhibition attenuates cardiac allograft remodeling secondary to down-regulation of M-TOR downstream targets and increased autophagy. There is a paucity of data regarding effect of Sirolimus, a M-TOR inhibitor, on human heart remodeling.

This aim of the proposal to identify the prevalence of cardiac allograft remodeling on current immunosuppressive strategies and determine risk factors for its development. It will also identify molecular pathways associated with cardiac allograft remodeling and determine the impact of Sirolimus on these pathways.

DETAILED DESCRIPTION:
Heart transplantation has become a well-established treatment option for patients with end-stage heart disease and currently has a one-year survival rate of 90%, a five-year survival rate of 70%, and 10-year survival rate of 50%. The introduction of anti-rejection treatment thirty years ago with drugs known as calcineurin inhibitors have resulted in a significant improvement in the survival of heart transplant recipients. However, most of this improvement occurs during the first year after transplantation. Beyond the first year, the mortality rate of heart transplant recipients has not changed, which indicates that the causes of late complications have not been affected in the last three decades by improvements in post-transplant care. It becomes apparent that in order to improve the late outcomes, the focus in heart transplant research needs to be shifted to the prevention and the treatment of late complications.

Cardiac allograft remodeling (CAR), or changes in heart's geometric pattern, is one of the common complications after heart transplantation and often inflicts poor quality of life, heart failure, and decreased survival. The risk factors and mechanism for the development and progression of CAR are poorly defined, and there is no effective treatment for this condition. In the proposed study, we will identify the prevalence, risk factors, and effect of CAR on physical capacity, cardiac vascular disease, and patient survival after a heart transplant. For assessment of heart geometry, we will use cardiac magnetic resonance imaging (CMRI), a techniques used to visualize the internal structures of the body in detail. CMRI is considered as being a "gold standard" for evaluating the heart's structure and function. We will also evaluate the molecular and genetic markers associated with development and progression of CAR after heart transplantation.

The drug Sirolimus, a new anti-rejection agent, can be used in place of calcineurin inhibitors after heart transplantation. Recent experimental and animal studies indicate that Sirolimus can attenuate the changes in the heart's geometry after a transplant (i.e., CAR) and improve heart function. We will assess the effect of Sirolimus on CAR in humans and will evaluate molecular and genetic markers associated with this effect.

It is our goal to provide an important insight into the nature of CAR after heart transplantation and its response to new anti-rejection drug Sirolimus. This information will have a significant impact on the treatment of heart transplant recipients and thus improve quality of life and prolong survival after heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All adult cardiac transplant recipients undergoing heart transplantation at UNMC/TNMC.

Exclusion Criteria:

* Adult cardiac transplant recipients with acute rejection (ISHLT R> grade 2) or acute infection.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Assessment in left ventricular hypertrophy | One year
  The primary end point will be the change from baseline in LV mass indexed to height in meters 2.7 and LV concentricity as assessed by MRI during 12 months of the treatment.

SECONDARY OUTCOMES:
Assess outcomes | One year
  The secondary end points will be changes from baseline in LV function.
Access outcomes | One year
  Exercise performance (peak VO2, equivalent for carbon dioxide (VE/VCO2)and coronary vessel intimal thickening.

OTHER OUTCOMES:
Safety end points | Three years
  Safety end points will be SRL side effects and prevalence of acute cellular cardiac rejection (ISHLT ≥ 2R) and AMR.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lowes, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Grossman E, Messerli FH. Hypertension and diabetes. Adv Cardiol. 2008;45:82-106. doi: 10.1159/000115189. PMID 18230957
- [Result] Levy D, Garrison RJ, Savage DD, Kannel WB, Castelli WP. Prognostic implications of echocardiographically determined left ventricular mass in the Framingham Heart Study. N Engl J Med. 1990 May 31;322(22):1561-6. doi: 10.1056/NEJM199005313222203. PMID 2139921
- [Result] Koren MJ, Devereux RB, Casale PN, Savage DD, Laragh JH. Relation of left ventricular mass and geometry to morbidity and mortality in uncomplicated essential hypertension. Ann Intern Med. 1991 Mar 1;114(5):345-52. doi: 10.7326/0003-4819-114-5-345. PMID 1825164
- [Result] Esposito G, Rapacciuolo A, Naga Prasad SV, Rockman HA. Cardiac hypertrophy: role of G protein-coupled receptors. J Card Fail. 2002 Dec;8(6 Suppl):S409-14. doi: 10.1054/jcaf.2002.129283. PMID 12555153
- [Result] Goodroe R, Bonnema DD, Lunsford S, Anderson P, Ryan-Baille B, Uber W, Ikonomidis J, Crumbley AJ, VanBakel A, Zile MR, Pereira N. Severe left ventricular hypertrophy 1 year after transplant predicts mortality in cardiac transplant recipients. J Heart Lung Transplant. 2007 Feb;26(2):145-51. doi: 10.1016/j.healun.2006.11.003. PMID 17258148
- [Result] Tischler MD, Lee RT, Plappert T, Mudge GH, St John Sutton M, Parker JD. Serial assessment of left ventricular function and mass after orthotopic heart transplantation: a 4-year longitudinal study. J Am Coll Cardiol. 1992 Jan;19(1):60-6. doi: 10.1016/0735-1097(92)90052-o. PMID 1729347
- [Result] Vigneswaran WT, Rumberger JA, Rodeheffer RJ, Breen JF, McGregor CG. Ventricular remodeling after orthotopic cardiac transplantation. Mayo Clin Proc. 1996 Aug;71(8):735-42. doi: 10.4065/71.8.735. PMID 8691893
- [Result] Raichlin E, Villarraga HR, Chandrasekaran K, Clavell AL, Frantz RP, Kushwaha SS, Rodeheffer RJ, McGregor CG, Daly RC, Park SJ, Kremers WK, Edwards BS, Pereira NL. Cardiac allograft remodeling after heart transplantation is associated with increased graft vasculopathy and mortality. Am J Transplant. 2009 Jan;9(1):132-9. doi: 10.1111/j.1600-6143.2008.02474.x. Epub 2008 Nov 27. PMID 19067662
- [Result] Hosenpud JD, Norman DJ, Cobanoglu MA, Floten HS, Conner RM, Starr A. Serial echocardiographic findings early after heart transplantation: evidence for reversible right ventricular dysfunction and myocardial edema. J Heart Transplant. 1987 Nov-Dec;6(6):343-7. PMID 2961856
- [Result] Raichlin E, Al-Omari MA, Hayes CL, Edwards BS, Frantz RP, Boilson BA, Clavell AL, Rodeheffer RJ, Schirger JA, Kushwaha SS, Allison TG, Pereira NL. Cardiac allograft hypertrophy is associated with impaired exercise tolerance after heart transplantation. J Heart Lung Transplant. 2011 Oct;30(10):1153-60. doi: 10.1016/j.healun.2011.04.012. Epub 2011 May 31. PMID 21621424
- [Result] Doggrell SA. Is everolimus useful in preventing allograft rejection and vasculopathy after heart transplant? Expert Opin Investig Drugs. 2004 Feb;13(2):161-3. doi: 10.1517/13543784.13.2.161. PMID 14996650
- [Result] Mancini D, Pinney S, Burkhoff D, LaManca J, Itescu S, Burke E, Edwards N, Oz M, Marks AR. Use of rapamycin slows progression of cardiac transplantation vasculopathy. Circulation. 2003 Jul 8;108(1):48-53. doi: 10.1161/01.CIR.0000070421.38604.2B. Epub 2003 May 12. PMID 12742978
- [Result] Raichlin E, Bae JH, Khalpey Z, Edwards BS, Kremers WK, Clavell AL, Rodeheffer RJ, Frantz RP, Rihal C, Lerman A, Kushwaha SS. Conversion to sirolimus as primary immunosuppression attenuates the progression of allograft vasculopathy after cardiac transplantation. Circulation. 2007 Dec 4;116(23):2726-33. doi: 10.1161/CIRCULATIONAHA.107.692996. Epub 2007 Nov 19. PMID 18025531
- [Result] Raichlin E, Edwards BS, Kremers WK, Clavell AL, Rodeheffer RJ, Frantz RP, Pereira NL, Daly RC, McGregor CG, Lerman A, Kushwaha SS. Acute cellular rejection and the subsequent development of allograft vasculopathy after cardiac transplantation. J Heart Lung Transplant. 2009 Apr;28(4):320-7. doi: 10.1016/j.healun.2009.01.006. PMID 19332257
- [Result] Patel PC, Reimold SC, Araj FG, Ayers CR, Kaiser PA, Peshock RM, Yancy CW, Ring WS, Gupta S, Mishkin JD, Mammen PP, Markham DW, Drazner MH. Concentric left ventricular hypertrophy as assessed by cardiac magnetic resonance imaging and risk of death in cardiac transplant recipients. J Heart Lung Transplant. 2010 Dec;29(12):1369-79. doi: 10.1016/j.healun.2010.05.008. PMID 20599402
- [Result] Kuppahally SS, Valantine HA, Weisshaar D, Parekh H, Hung YY, Haddad F, Fowler M, Vagelos R, Perlroth MG, Robbins RC, Hunt SA. Outcome in cardiac recipients of donor hearts with increased left ventricular wall thickness. Am J Transplant. 2007 Oct;7(10):2388-95. doi: 10.1111/j.1600-6143.2007.01930.x. PMID 17845572
- [Result] Stewart S, Winters GL, Fishbein MC, Tazelaar HD, Kobashigawa J, Abrams J, Andersen CB, Angelini A, Berry GJ, Burke MM, Demetris AJ, Hammond E, Itescu S, Marboe CC, McManus B, Reed EF, Reinsmoen NL, Rodriguez ER, Rose AG, Rose M, Suciu-Focia N, Zeevi A, Billingham ME. Revision of the 1990 working formulation for the standardization of nomenclature in the diagnosis of heart rejection. J Heart Lung Transplant. 2005 Nov;24(11):1710-20. doi: 10.1016/j.healun.2005.03.019. Epub 2005 Jun 20. PMID 16297770
- [Result] Billingham M, Kobashigawa JA. The revised ISHLT heart biopsy grading scale. J Heart Lung Transplant. 2005 Nov;24(11):1709. doi: 10.1016/j.healun.2005.03.018. No abstract available. PMID 16297769
- [Result] Grattan MT, Moreno-Cabral CE, Starnes VA, Oyer PE, Stinson EB, Shumway NE. Eight-year results of cyclosporine-treated patients with cardiac transplants. J Thorac Cardiovasc Surg. 1990 Mar;99(3):500-9. PMID 2308368
- [Result] Lemstrom K, Sihvola R, Bruggeman C, Hayry P, Koskinen P. Cytomegalovirus infection-enhanced cardiac allograft vasculopathy is abolished by DHPG prophylaxis in the rat. Circulation. 1997 Jun 17;95(12):2614-6. doi: 10.1161/01.cir.95.12.2614. PMID 9193428
- [Result] McDonald K, Rector TS, Braulin EA, Kubo SH, Olivari MT. Association of coronary artery disease in cardiac transplant recipients with cytomegalovirus infection. Am J Cardiol. 1989 Aug 1;64(5):359-62. doi: 10.1016/0002-9149(89)90535-3. PMID 2547298
- [Result] Peura JL, Zile MR, Feldman DS, VanBakel AB, McClure C, Uber W, Haynes H, Pereira NL. Effects of conversion from cyclosporine to tacrolimus on left ventricular structure in cardiac allograft recipients. J Heart Lung Transplant. 2005 Nov;24(11):1969-72. doi: 10.1016/j.healun.2005.02.011. PMID 16297806
- [Result] Karch SB, Billingham ME. Cyclosporine induced myocardial fibrosis: a unique controlled case report. J Heart Transplant. 1985 Feb;4(2):210-2. PMID 3916487
- [Result] Aziz S, Soine LA, Lewis SL, Kruse AP, Levy WC, Wehe KM, Fishbien DP, Allen MD. Donor left ventricular hypertrophy increases risk for early graft failure. Transpl Int. 1997;10(6):446-50. doi: 10.1007/s001470050084. PMID 9428118
- [Result] Lips DJ, deWindt LJ, van Kraaij DJ, Doevendans PA. Molecular determinants of myocardial hypertrophy and failure: alternative pathways for beneficial and maladaptive hypertrophy. Eur Heart J. 2003 May;24(10):883-96. doi: 10.1016/s0195-668x(02)00829-1. PMID 12714020
- [Result] Molkentin JD, Lu JR, Antos CL, Markham B, Richardson J, Robbins J, Grant SR, Olson EN. A calcineurin-dependent transcriptional pathway for cardiac hypertrophy. Cell. 1998 Apr 17;93(2):215-28. doi: 10.1016/s0092-8674(00)81573-1. PMID 9568714
- [Result] Malik FS, Mehra MR, Ventura HO, Smart FW, Stapleton DD, Ochsner JL. Management of cardiac allograft vasculopathy by transmyocardial laser revascularization. Am J Cardiol. 1997 Jul 15;80(2):224-5. doi: 10.1016/s0002-9149(97)00327-5. PMID 9230169
- [Result] Costanzo MR, Naftel DC, Pritzker MR, Heilman JK 3rd, Boehmer JP, Brozena SC, Dec GW, Ventura HO, Kirklin JK, Bourge RC, Miller LW. Heart transplant coronary artery disease detected by coronary angiography: a multiinstitutional study of preoperative donor and recipient risk factors. Cardiac Transplant Research Database. J Heart Lung Transplant. 1998 Aug;17(8):744-53. PMID 9730422
- [Result] Schwitter J, Saeed M, Wendland MF, Sakuma H, Bremerich J, Canet E, Higgins CB. Assessment of myocardial function and perfusion in a canine model of non-occlusive coronary artery stenosis using fast magnetic resonance imaging. J Magn Reson Imaging. 1999 Jan;9(1):101-10. doi: 10.1002/(sici)1522-2586(199901)9:13.0.co;2-9. PMID 10030657
- [Result] Khanna AK, Cairns VR, Becker CG, Hosenpud JD. Transforming growth factor (TGF)-beta mimics and anti-TGF-beta antibody abrogates the in vivo effects of cyclosporine: demonstration of a direct role of TGF-beta in immunosuppression and nephrotoxicity of cyclosporine. Transplantation. 1999 Mar 27;67(6):882-9. doi: 10.1097/00007890-199903270-00016. PMID 10199738
- [Result] Hojo M, Morimoto T, Maluccio M, Asano T, Morimoto K, Lagman M, Shimbo T, Suthanthiran M. Cyclosporine induces cancer progression by a cell-autonomous mechanism. Nature. 1999 Feb 11;397(6719):530-4. doi: 10.1038/17401. PMID 10028970
- [Result] Zhang D, Gaussin V, Taffet GE, Belaguli NS, Yamada M, Schwartz RJ, Michael LH, Overbeek PA, Schneider MD. TAK1 is activated in the myocardium after pressure overload and is sufficient to provoke heart failure in transgenic mice. Nat Med. 2000 May;6(5):556-63. doi: 10.1038/75037. PMID 10802712
- [Result] Feeley BT, Park AK, Hoyt EG, Robbins RC. Sulfasalazine inhibits reperfusion injury and prolongs allograft survival in rat cardiac transplants. J Heart Lung Transplant. 1999 Nov;18(11):1088-95. doi: 10.1016/s1053-2498(99)00078-9. PMID 10598732
- [Result] Mijares A, Malecot CO, Peineau N, Argibay JA. In vivo and in vitro inhibition of the L-type calcium current in isolated guinea-pig cardiomyocytes by the immunosuppressive agent cyclosporin A. J Mol Cell Cardiol. 1997 Aug;29(8):2067-76. doi: 10.1006/jmcc.1997.0441. PMID 9281439
- [Result] Marx SO, Reiken S, Hisamatsu Y, Jayaraman T, Burkhoff D, Rosemblit N, Marks AR. PKA phosphorylation dissociates FKBP12.6 from the calcium release channel (ryanodine receptor): defective regulation in failing hearts. Cell. 2000 May 12;101(4):365-76. doi: 10.1016/s0092-8674(00)80847-8. PMID 10830164
- [Result] Globits S, De Marco T, Schwitter J, Sakuma H, O'Sullivan M, Rifkin C, Keith F, Chatterjee K, Parmley WW, Higgins CB. Assessment of early left ventricular remodeling in orthotopic heart transplant recipients with cine magnetic resonance imaging: potential mechanisms. J Heart Lung Transplant. 1997 May;16(5):504-10. PMID 9171268
- [Result] Chareonthaitawee P, Christian TF, Miller TD, Hodge DO, Gibbons RJ. Correlation of resting first-pass left ventricular ejection fraction and resting myocardial infarct size. Am J Cardiol. 1998 Jun 1;81(11):1281-5. doi: 10.1016/s0002-9149(98)00156-8. PMID 9631963
- [Result] Espino G, Denney J, Furlong T, Fitzsimmons W, Nash RA. Assessment of myocardial hypertrophy by echocardiography in adult patients receiving tacrolimus or cyclosporine therapy for prevention of acute GVHD. Bone Marrow Transplant. 2001 Dec;28(12):1097-103. doi: 10.1038/sj.bmt.1703304. PMID 11803349
- [Result] Atkison P, Joubert G, Barron A, Grant D, Paradis K, Seidman E, Wall W, Rosenberg H, Howard J, Williams S, et al. Hypertrophic cardiomyopathy associated with tacrolimus in paediatric transplant patients. Lancet. 1995 Apr 8;345(8954):894-6. doi: 10.1016/s0140-6736(95)90011-x. PMID 7535875
- [Result] Kushwaha SS, Raichlin E, Sheinin Y, Kremers WK, Chandrasekaran K, Brunn GJ, Platt JL. Sirolimus affects cardiomyocytes to reduce left ventricular mass in heart transplant recipients. Eur Heart J. 2008 Nov;29(22):2742-50. doi: 10.1093/eurheartj/ehn407. Epub 2008 Sep 11. PMID 18790727
- [Result] Frey N, Barrientos T, Shelton JM, Frank D, Rutten H, Gehring D, Kuhn C, Lutz M, Rothermel B, Bassel-Duby R, Richardson JA, Katus HA, Hill JA, Olson EN. Mice lacking calsarcin-1 are sensitized to calcineurin signaling and show accelerated cardiomyopathy in response to pathological biomechanical stress. Nat Med. 2004 Dec;10(12):1336-43. doi: 10.1038/nm1132. Epub 2004 Nov 14. PMID 15543153
- [Result] Armstrong AT, Binkley PF, Baker PB, Myerowitz PD, Leier CV. Quantitative investigation of cardiomyocyte hypertrophy and myocardial fibrosis over 6 years after cardiac transplantation. J Am Coll Cardiol. 1998 Sep;32(3):704-10. doi: 10.1016/s0735-1097(98)00296-4. PMID 9741515
- [Result] Rouleau JL, de Champlain J, Klein M, Bichet D, Moye L, Packer M, Dagenais GR, Sussex B, Arnold JM, Sestier F, et al. Activation of neurohumoral systems in postinfarction left ventricular dysfunction. J Am Coll Cardiol. 1993 Aug;22(2):390-8. doi: 10.1016/0735-1097(93)90042-y. PMID 8101532
- [Result] Soonpaa MH, Kim KK, Pajak L, Franklin M, Field LJ. Cardiomyocyte DNA synthesis and binucleation during murine development. Am J Physiol. 1996 Nov;271(5 Pt 2):H2183-9. doi: 10.1152/ajpheart.1996.271.5.H2183. PMID 8945939
- [Result] McGill CJ, Brooks G. Cell cycle control mechanisms and their role in cardiac growth. Cardiovasc Res. 1995 Oct;30(4):557-69. No abstract available. PMID 8575004
- [Result] Brooks G, Poolman RA, McGill CJ, Li JM. Expression and activities of cyclins and cyclin-dependent kinases in developing rat ventricular myocytes. J Mol Cell Cardiol. 1997 Aug;29(8):2261-71. doi: 10.1006/jmcc.1997.0471. PMID 9281457
- [Result] Poolman RA, Gilchrist R, Brooks G. Cell cycle profiles and expressions of p21CIP1 AND P27KIP1 during myocyte development. Int J Cardiol. 1998 Dec 1;67(2):133-42. doi: 10.1016/s0167-5273(98)00320-9. PMID 9891946
- [Result] Capasso JM, Bruno S, Cheng W, Li P, Rodgers R, Darzynkiewicz Z, Anversa P. Ventricular loading is coupled with DNA synthesis in adult cardiac myocytes after acute and chronic myocardial infarction in rats. Circ Res. 1992 Dec;71(6):1379-89. doi: 10.1161/01.res.71.6.1379. PMID 1423934
- [Result] Hannan KM, Brandenburger Y, Jenkins A, Sharkey K, Cavanaugh A, Rothblum L, Moss T, Poortinga G, McArthur GA, Pearson RB, Hannan RD. mTOR-dependent regulation of ribosomal gene transcription requires S6K1 and is mediated by phosphorylation of the carboxy-terminal activation domain of the nucleolar transcription factor UBF. Mol Cell Biol. 2003 Dec;23(23):8862-77. doi: 10.1128/MCB.23.23.8862-8877.2003. PMID 14612424
- [Result] Molkentin JD. Calcineurin and beyond: cardiac hypertrophic signaling. Circ Res. 2000 Oct 27;87(9):731-8. doi: 10.1161/01.res.87.9.731. PMID 11055975
- [Result] Schmelzle T, Hall MN. TOR, a central controller of cell growth. Cell. 2000 Oct 13;103(2):253-62. doi: 10.1016/s0092-8674(00)00117-3. PMID 11057898
- [Result] Sehgal SN, Czerkawski H, Kudelski A, Pandev K, Saucier R, Vezina C. Ravidomycin (AY-25,545), a new antitumor antibiotic. J Antibiot (Tokyo). 1983 Apr;36(4):355-61. doi: 10.7164/antibiotics.36.355. PMID 6853365
- [Result] Marx SO, Marks AR. Bench to bedside: the development of rapamycin and its application to stent restenosis. Circulation. 2001 Aug 21;104(8):852-5. doi: 10.1161/01.cir.104.8.852. No abstract available. PMID 11514367
- [Result] Kushwaha SS, Khalpey Z, Frantz RP, Rodeheffer RJ, Clavell AL, Daly RC, McGregor CG, Edwards BS. Sirolimus in cardiac transplantation: use as a primary immunosuppressant in calcineurin inhibitor-induced nephrotoxicity. J Heart Lung Transplant. 2005 Dec;24(12):2129-36. doi: 10.1016/j.healun.2005.08.015. PMID 16364861
- [Result] Hausleiter J, Kastrati A, Mehilli J, Vogeser M, Zohlnhofer D, Schuhlen H, Goos C, Pache J, Dotzer F, Pogatsa-Murray G, Dirschinger J, Heemann U, Schomig A; OSIRIS Investigators. Randomized, double-blind, placebo-controlled trial of oral sirolimus for restenosis prevention in patients with in-stent restenosis: the Oral Sirolimus to Inhibit Recurrent In-stent Stenosis (OSIRIS) trial. Circulation. 2004 Aug 17;110(7):790-5. doi: 10.1161/01.CIR.0000138935.17503.35. Epub 2004 Aug 9. PMID 15302787
- [Result] McMullen JR, Shioi T, Zhang L, Tarnavski O, Sherwood MC, Dorfman AL, Longnus S, Pende M, Martin KA, Blenis J, Thomas G, Izumo S. Deletion of ribosomal S6 kinases does not attenuate pathological, physiological, or insulin-like growth factor 1 receptor-phosphoinositide 3-kinase-induced cardiac hypertrophy. Mol Cell Biol. 2004 Jul;24(14):6231-40. doi: 10.1128/MCB.24.14.6231-6240.2004. PMID 15226426
- [Result] Shioi T, McMullen JR, Tarnavski O, Converso K, Sherwood MC, Manning WJ, Izumo S. Rapamycin attenuates load-induced cardiac hypertrophy in mice. Circulation. 2003 Apr 1;107(12):1664-70. doi: 10.1161/01.CIR.0000057979.36322.88. Epub 2003 Mar 17. PMID 12668503
- [Result] Buss SJ, Muenz S, Riffel JH, Malekar P, Hagenmueller M, Weiss CS, Bea F, Bekeredjian R, Schinke-Braun M, Izumo S, Katus HA, Hardt SE. Beneficial effects of Mammalian target of rapamycin inhibition on left ventricular remodeling after myocardial infarction. J Am Coll Cardiol. 2009 Dec 15;54(25):2435-46. doi: 10.1016/j.jacc.2009.08.031. PMID 20082935
- [Result] Li JM, Brooks G. Cell cycle regulatory molecules (cyclins, cyclin-dependent kinases and cyclin-dependent kinase inhibitors) and the cardiovascular system; potential targets for therapy? Eur Heart J. 1999 Mar;20(6):406-20. doi: 10.1053/euhj.1998.1308. PMID 10213344
- [Result] Nourse J, Firpo E, Flanagan WM, Coats S, Polyak K, Lee MH, Massague J, Crabtree GR, Roberts JM. Interleukin-2-mediated elimination of the p27Kip1 cyclin-dependent kinase inhibitor prevented by rapamycin. Nature. 1994 Dec 8;372(6506):570-3. doi: 10.1038/372570a0. PMID 7990932
- [Result] Nakayama K, Ishida N, Shirane M, Inomata A, Inoue T, Shishido N, Horii I, Loh DY, Nakayama K. Mice lacking p27(Kip1) display increased body size, multiple organ hyperplasia, retinal dysplasia, and pituitary tumors. Cell. 1996 May 31;85(5):707-20. doi: 10.1016/s0092-8674(00)81237-4. PMID 8646779
- [Result] Hauck L, Harms C, An J, Rohne J, Gertz K, Dietz R, Endres M, von Harsdorf R. Protein kinase CK2 links extracellular growth factor signaling with the control of p27(Kip1) stability in the heart. Nat Med. 2008 Mar;14(3):315-24. doi: 10.1038/nm1729. Epub 2008 Mar 2. PMID 18311148
- [Result] Kato JY, Matsuoka M, Polyak K, Massague J, Sherr CJ. Cyclic AMP-induced G1 phase arrest mediated by an inhibitor (p27Kip1) of cyclin-dependent kinase 4 activation. Cell. 1994 Nov 4;79(3):487-96. doi: 10.1016/0092-8674(94)90257-7. PMID 7954814
- [Result] Kitsis RN, Peng CF, Cuervo AM. Eat your heart out. Nat Med. 2007 May;13(5):539-41. doi: 10.1038/nm0507-539. No abstract available. PMID 17479097
- [Result] Nakai A, Yamaguchi O, Takeda T, Higuchi Y, Hikoso S, Taniike M, Omiya S, Mizote I, Matsumura Y, Asahi M, Nishida K, Hori M, Mizushima N, Otsu K. The role of autophagy in cardiomyocytes in the basal state and in response to hemodynamic stress. Nat Med. 2007 May;13(5):619-24. doi: 10.1038/nm1574. Epub 2007 Apr 22. PMID 17450150
- [Result] Rubinsztein DC, Gestwicki JE, Murphy LO, Klionsky DJ. Potential therapeutic applications of autophagy. Nat Rev Drug Discov. 2007 Apr;6(4):304-12. doi: 10.1038/nrd2272. PMID 17396135
- [Result] Wang BT, Ducker GS, Barczak AJ, Barbeau R, Erle DJ, Shokat KM. The mammalian target of rapamycin regulates cholesterol biosynthetic gene expression and exhibits a rapamycin-resistant transcriptional profile. Proc Natl Acad Sci U S A. 2011 Sep 13;108(37):15201-6. doi: 10.1073/pnas.1103746108. Epub 2011 Aug 29. PMID 21876130
- [Result] Wang Z, Gerstein M, Snyder M. RNA-Seq: a revolutionary tool for transcriptomics. Nat Rev Genet. 2009 Jan;10(1):57-63. doi: 10.1038/nrg2484. PMID 19015660
- [Result] Missouris CG, Forbat SM, Singer DR, Markandu ND, Underwood R, MacGregor GA. Echocardiography overestimates left ventricular mass: a comparative study with magnetic resonance imaging in patients with hypertension. J Hypertens. 1996 Aug;14(8):1005-10. PMID 8884556
- [Result] Stewart GA, Foster J, Cowan M, Rooney E, McDonagh T, Dargie HJ, Rodger RS, Jardine AG. Echocardiography overestimates left ventricular mass in hemodialysis patients relative to magnetic resonance imaging. Kidney Int. 1999 Dec;56(6):2248-53. doi: 10.1046/j.1523-1755.1999.00786.x. PMID 10594802
- [Result] Hedeer F, Palmer J, Arheden H, Ugander M. Gated myocardial perfusion SPECT underestimates left ventricular volumes and shows high variability compared to cardiac magnetic resonance imaging -- a comparison of four different commercial automated software packages. BMC Med Imaging. 2010 May 25;10:10. doi: 10.1186/1471-2342-10-10. PMID 20500866
- [Result] Harel F, Finnerty V, Gregoire J, Thibault B, Marcotte F, Ugolini P, Khairy P. Gated blood-pool SPECT versus cardiac magnetic resonance imaging for the assessment of left ventricular volumes and ejection fraction. J Nucl Cardiol. 2010 Jun;17(3):427-34. doi: 10.1007/s12350-010-9195-5. Epub 2010 Feb 12. PMID 20151236
- [Result] Bellenger NG, Burgess MI, Ray SG, Lahiri A, Coats AJ, Cleland JG, Pennell DJ. Comparison of left ventricular ejection fraction and volumes in heart failure by echocardiography, radionuclide ventriculography and cardiovascular magnetic resonance; are they interchangeable? Eur Heart J. 2000 Aug;21(16):1387-96. doi: 10.1053/euhj.2000.2011. PMID 10952828
- [Result] Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol. 2002 Jul 1;90(1):29-34. doi: 10.1016/s0002-9149(02)02381-0. PMID 12088775
- [Result] Ciliberto GR, Mascarello M, Gronda E, Bonacina E, Anjos MC, Danzi G, Colombo P, Frigerio M, Alberti A, De Vita C. Acute rejection after heart transplantation: noninvasive echocardiographic evaluation. J Am Coll Cardiol. 1994 Apr;23(5):1156-61. doi: 10.1016/0735-1097(94)90605-x. PMID 8144783
- [Result] Hudsmith LE, Petersen SE, Tyler DJ, Francis JM, Cheng AS, Clarke K, Selvanayagam JB, Robson MD, Neubauer S. Determination of cardiac volumes and mass with FLASH and SSFP cine sequences at 1.5 vs. 3 Tesla: a validation study. J Magn Reson Imaging. 2006 Aug;24(2):312-8. doi: 10.1002/jmri.20638. PMID 16795076
- [Result] Malayeri AA, Johnson WC, Macedo R, Bathon J, Lima JA, Bluemke DA. Cardiac cine MRI: Quantification of the relationship between fast gradient echo and steady-state free precession for determination of myocardial mass and volumes. J Magn Reson Imaging. 2008 Jul;28(1):60-6. doi: 10.1002/jmri.21405. PMID 18581356
- [Result] Carlsson M, Ubachs JF, Hedstrom E, Heiberg E, Jovinge S, Arheden H. Myocardium at risk after acute infarction in humans on cardiac magnetic resonance: quantitative assessment during follow-up and validation with single-photon emission computed tomography. JACC Cardiovasc Imaging. 2009 May;2(5):569-76. doi: 10.1016/j.jcmg.2008.11.018. PMID 19442942
- [Result] Gallo P, Baroldi G, Thiene G, Agozzino L, Arbustini E, Bartoloni G, Bonacina E, Bosman C, Catani G, Cocco P, et al. When and why do heart transplant recipients die? A 7 year experience of 1068 cardiac transplants. Virchows Arch A Pathol Anat Histopathol. 1993;422(6):453-8. doi: 10.1007/BF01606453. PMID 8333149
- [Result] Almenar L, Igual B, Martinez-Dolz L, Arnau MA, Osa A, Rueda J, Palencia M. Utility of cardiac magnetic resonance imaging for the diagnosis of heart transplant rejection. Transplant Proc. 2003 Aug;35(5):1962-4. doi: 10.1016/s0041-1345(03)00653-5. PMID 12962864
- [Result] Aherne T, Tscholakoff D, Finkbeiner W, Sechtem U, Derugin N, Yee E, Higgins CB. Magnetic resonance imaging of cardiac transplants: the evaluation of rejection of cardiac allografts with and without immunosuppression. Circulation. 1986 Jul;74(1):145-56. doi: 10.1161/01.cir.74.1.145. PMID 3518982
- [Result] Marie PY, Carteaux JP, Escanye JM, Claudon O, David N, Mattei S, Hassan N, Danchin N, Karcher G, Bertrand A, Villemot JP. Detection and prediction of acute heart transplant rejection with the myocardial T2 determination provided by a black-blood magnetic resonance imaging sequence. J Heart Lung Transplant. 2001 Feb;20(2):193-194. doi: 10.1016/s1053-2498(00)00406-x. No abstract available. PMID 11250334
- [Result] Giri S, Chung YC, Merchant A, Mihai G, Rajagopalan S, Raman SV, Simonetti OP. T2 quantification for improved detection of myocardial edema. J Cardiovasc Magn Reson. 2009 Dec 30;11(1):56. doi: 10.1186/1532-429X-11-56. PMID 20042111
- [Result] Lund G, Morin RL, Olivari MT, Ring WS. Serial myocardial T2 relaxation time measurements in normal subjects and heart transplant recipients. J Heart Transplant. 1988 Jul-Aug;7(4):274-9. PMID 2845037
- [Result] Rudolph A, Abdel-Aty H, Bohl S, Boye P, Zagrosek A, Dietz R, Schulz-Menger J. Noninvasive detection of fibrosis applying contrast-enhanced cardiac magnetic resonance in different forms of left ventricular hypertrophy relation to remodeling. J Am Coll Cardiol. 2009 Jan 20;53(3):284-91. doi: 10.1016/j.jacc.2008.08.064. PMID 19147047
- [Result] Schulz-Menger J, Gross M, Messroghli D, Uhlich F, Dietz R, Friedrich MG. Cardiovascular magnetic resonance of acute myocardial infarction at a very early stage. J Am Coll Cardiol. 2003 Aug 6;42(3):513-8. doi: 10.1016/s0735-1097(03)00717-4. PMID 12906982
- [Result] Kim RJ, Fieno DS, Parrish TB, Harris K, Chen EL, Simonetti O, Bundy J, Finn JP, Klocke FJ, Judd RM. Relationship of MRI delayed contrast enhancement to irreversible injury, infarct age, and contractile function. Circulation. 1999 Nov 9;100(19):1992-2002. doi: 10.1161/01.cir.100.19.1992. PMID 10556226
- [Result] Patel MR, Cawley PJ, Heitner JF, Klem I, Parker MA, Jaroudi WA, Meine TJ, White JB, Elliott MD, Kim HW, Judd RM, Kim RJ. Detection of myocardial damage in patients with sarcoidosis. Circulation. 2009 Nov 17;120(20):1969-77. doi: 10.1161/CIRCULATIONAHA.109.851352. Epub 2009 Nov 2. PMID 19884472
- [Result] Steen H, Merten C, Refle S, Klingenberg R, Dengler T, Giannitsis E, Katus HA. Prevalence of different gadolinium enhancement patterns in patients after heart transplantation. J Am Coll Cardiol. 2008 Sep 30;52(14):1160-7. doi: 10.1016/j.jacc.2008.05.059. PMID 18804744
- [Result] Grady KL. Quality of life after heart transplantation: are things really better? Curr Opin Cardiol. 2003 Mar;18(2):129-35. doi: 10.1097/00001573-200303000-00011. PMID 12652219
- [Result] Osada N, Chaitman BR, Donohue TJ, Wolford TL, Stelken AM, Miller LW. Long-term cardiopulmonary exercise performance after heart transplantation. Am J Cardiol. 1997 Feb 15;79(4):451-6. doi: 10.1016/s0002-9149(96)00785-0. PMID 9052349
- [Result] Raichlin E, Chandrasekaran K, Kremers WK, Frantz RP, Clavell AL, Pereira NL, Rodeheffer RJ, Daly RC, McGregor CG, Edwards BS, Kushwaha SS. Sirolimus as primary immunosuppressant reduces left ventricular mass and improves diastolic function of the cardiac allograft. Transplantation. 2008 Nov 27;86(10):1395-400. doi: 10.1097/TP.0b013e318189049a. PMID 19034009
- [Result] de Simone G, Daniels SR, Kimball TR, Roman MJ, Romano C, Chinali M, Galderisi M, Devereux RB. Evaluation of concentric left ventricular geometry in humans: evidence for age-related systematic underestimation. Hypertension. 2005 Jan;45(1):64-8. doi: 10.1161/01.HYP.0000150108.37527.57. Epub 2004 Nov 22. PMID 15557389
- [Result] Bae JH, Rihal CS, Edwards BS, Kushwaha SS, Mathew V, Prasad A, Holmes DR Jr, Lerman A. Association of angiotensin-converting enzyme inhibitors and serum lipids with plaque regression in cardiac allograft vasculopathy. Transplantation. 2006 Oct 27;82(8):1108-11. doi: 10.1097/01.tp.0000230378.61437.a5. PMID 17060862
- [Result] Chaves AJ, Sousa AG, Mattos LA, Abizaid A, Staico R, Feres F, Centemero M, Tanajura LF, Abizaid A, Pinto I, Maldonado G, Seixas A, Costa MA, Paes A, Mintz GS, Sousa JE. Volumetric analysis of in-stent intimal hyperplasia in diabetic patients treated with or without abciximab: results of the Diabetes Abciximab steNT Evaluation (DANTE) randomized trial. Circulation. 2004 Feb 24;109(7):861-6. doi: 10.1161/01.CIR.0000116752.12261.D4. Epub 2004 Feb 2. PMID 14757690
- [Result] Daida H, Allison TG, Johnson BD, Squires RW, Gau GT. Further increase in oxygen uptake during early active recovery following maximal exercise in chronic heart failure. Chest. 1996 Jan;109(1):47-51. doi: 10.1378/chest.109.1.47. PMID 8549215
- [Result] Ross RM. ATS/ACCP statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 May 15;167(10):1451; author reply 1451. doi: 10.1164/ajrccm.167.10.950. No abstract available. PMID 12738602
- [Result] Nagalakshmi U, Wang Z, Waern K, Shou C, Raha D, Gerstein M, Snyder M. The transcriptional landscape of the yeast genome defined by RNA sequencing. Science. 2008 Jun 6;320(5881):1344-9. doi: 10.1126/science.1158441. Epub 2008 May 1. PMID 18451266
- [Result] Lowes BD, Baker ML, Blaxall BC. Gene expression profile of the recovering human heart. Eur Heart J. 2007 Mar;28(5):522-4. doi: 10.1093/eurheartj/ehl555. Epub 2007 Feb 21. No abstract available. PMID 17314109
- [Result] Heinze G, Puhr R. Bias-reduced and separation-proof conditional logistic regression with small or sparse data sets. Stat Med. 2010 Mar 30;29(7-8):770-7. doi: 10.1002/sim.3794. PMID 20213709
- [Result] Costanzo MR, Dipchand A, Starling R, Anderson A, Chan M, Desai S, Fedson S, Fisher P, Gonzales-Stawinski G, Martinelli L, McGiffin D, Smith J, Taylor D, Meiser B, Webber S, Baran D, Carboni M, Dengler T, Feldman D, Frigerio M, Kfoury A, Kim D, Kobashigawa J, Shullo M, Stehlik J, Teuteberg J, Uber P, Zuckermann A, Hunt S, Burch M, Bhat G, Canter C, Chinnock R, Crespo-Leiro M, Delgado R, Dobbels F, Grady K, Kao W, Lamour J, Parry G, Patel J, Pini D, Towbin J, Wolfel G, Delgado D, Eisen H, Goldberg L, Hosenpud J, Johnson M, Keogh A, Lewis C, O'Connell J, Rogers J, Ross H, Russell S, Vanhaecke J; International Society of Heart and Lung Transplantation Guidelines. The International Society of Heart and Lung Transplantation Guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2010 Aug;29(8):914-56. doi: 10.1016/j.healun.2010.05.034. No abstract available. PMID 20643330
- [Result] Dean PG, Lund WJ, Larson TS, Prieto M, Nyberg SL, Ishitani MB, Kremers WK, Stegall MD. Wound-healing complications after kidney transplantation: a prospective, randomized comparison of sirolimus and tacrolimus. Transplantation. 2004 May 27;77(10):1555-61. doi: 10.1097/01.tp.0000123082.31092.53. PMID 15239621
- [Result] Kuppahally S, Al-Khaldi A, Weisshaar D, Valantine HA, Oyer P, Robbins RC, Hunt SA. Wound healing complications with de novo sirolimus versus mycophenolate mofetil-based regimen in cardiac transplant recipients. Am J Transplant. 2006 May;6(5 Pt 1):986-92. doi: 10.1111/j.1600-6143.2006.01282.x. PMID 16611334
- [Result] Trapnell C, Williams BA, Pertea G, Mortazavi A, Kwan G, van Baren MJ, Salzberg SL, Wold BJ, Pachter L. Transcript assembly and quantification by RNA-Seq reveals unannotated transcripts and isoform switching during cell differentiation. Nat Biotechnol. 2010 May;28(5):511-5. doi: 10.1038/nbt.1621. Epub 2010 May 2. PMID 20436464
- [Result] Trapnell C, Pachter L, Salzberg SL. TopHat: discovering splice junctions with RNA-Seq. Bioinformatics. 2009 May 1;25(9):1105-11. doi: 10.1093/bioinformatics/btp120. Epub 2009 Mar 16. PMID 19289445
- [Result] Langmead B, Trapnell C, Pop M, Salzberg SL. Ultrafast and memory-efficient alignment of short DNA sequences to the human genome. Genome Biol. 2009;10(3):R25. doi: 10.1186/gb-2009-10-3-r25. Epub 2009 Mar 4. PMID 19261174
- [Result] Goecks J, Nekrutenko A, Taylor J; Galaxy Team. Galaxy: a comprehensive approach for supporting accessible, reproducible, and transparent computational research in the life sciences. Genome Biol. 2010;11(8):R86. doi: 10.1186/gb-2010-11-8-r86. Epub 2010 Aug 25. PMID 20738864
- [Result] Reich M, Liefeld T, Gould J, Lerner J, Tamayo P, Mesirov JP. GenePattern 2.0. Nat Genet. 2006 May;38(5):500-1. doi: 10.1038/ng0506-500. No abstract available. PMID 16642009
- [Result] Nosal WH, Thompson DW, Yan L, Sarkar S, Subramanian A, Woollam JA. Infrared optical properties and AFM of spin-cast chitosan films chemically modified with 1,2 Epoxy-3-phenoxy-propane. Colloids Surf B Biointerfaces. 2005 Nov 25;46(1):26-31. doi: 10.1016/j.colsurfb.2005.08.006. Epub 2005 Sep 30. PMID 16199143
- [Result] Li J, Witten DM, Johnstone IM, Tibshirani R. Normalization, testing, and false discovery rate estimation for RNA-sequencing data. Biostatistics. 2012 Jul;13(3):523-38. doi: 10.1093/biostatistics/kxr031. Epub 2011 Oct 14. PMID 22003245